CLINICAL TRIAL: NCT00282854
Title: Genetics of Rolandic Epilepsy
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4727; R01NS047530 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2011-08

CONDITIONS: Epilepsy
Keywords: epilepsy; Rolandic epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsy, Rolandic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: Cases: Children with rolandic epilepsy
- Group II: Controls: Individuals group matched to cases for ethnicity, sex and area of residence but lacking a primary brain disorder.

SUMMARY:
The purpose of this study is to find the genes that cause Rolandic epilepsy and its related traits.

DETAILED DESCRIPTION:
Rolandic epilepsy (RE) is the most common type of childhood epilepsy-affecting more than 50,000 children in the United States-and has a complex genetic inheritance. The seizure prognosis is relatively benign, however, many children with RE also have problems with speech and language, reading, and motor coordination. Symptoms of the disorder overlap with more severe types of epilepsy.

The purpose of this study is to find the genes that influence RE and its related traits. Identifying genetic causes for the variants would improve diagnosis and allow for early intervention.

Researchers will enroll 1000 children with RE and 3000 controls for participation in the study. The scientists will request medical histories and (salivary) DNA samples from the participants. Participation can be completed by mail and telephone.

Results from this study should provide important information regarding diagnosis and prognosis of RE, may be useful in clinical management, and, eventually, may lead to a cure for this and other forms of epilepsy.

ELIGIBILITY:
Inclusion:

* typical history of focal seizures
* EEG centrotemporal sharp waves
* age of onset 3-12 years
* no previous epilepsy type (febrile seizures OK)
* normal development
* normal neurological examination
* normal MRI/CT (if done)

Exclusion:

* only history of secondary generalized seizures
* atypical history/semiology
* history and EEG inconsistent
* abnormal EEG background
* very early (<3yrs) or late (>12yrs) onset
* global neurodevelopmental deficit
* deviant neurodevelopment
* structural imaging abnormality

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deb K. Pal, MD, PhD, Principal Investigator — Associate Research Scientist, Mailman School of Public Health, Columbia University Medical Center
Locations (1):
- Mailman School of Public Health, Columbia University Medical Center, 722 West 168th St, 6th Floor, New York, New York, United States

REFERENCES:
- See also: study website — http://www.rolandic.com